CLINICAL TRIAL: NCT05379036
Title: The Role of Intestinal Permeability and Intestinal Microbiota in the Development of the Irritable Bowel Syndrome and Functional Dyspepsia Symptoms
Brief Title: Intestinal Permeability and Intestinal Microbiota in Irritable Bowel Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 116227
Record Dates: First submitted 2022-03-31; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-03

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): a group of patients who, after the examination, were prescribed therapy with trimebutine 600 mg per day for 2 months
  Interventions: Drug: prescribing anapproved drug, examination
- Group B (Experimental): a group of patients who, after the examination, were prescribed therapy with rebamipide 300 mg per day for 2 months
  Interventions: Drug: prescribing anapproved drug, examination
- Group C (Experimental): a group of patients who, after the examination, were prescribed therapy with trimebutine 600 mg per day + rebamipide 300 mg per day for 2 months
  Interventions: Drug: prescribing anapproved drug, examination
- Control (No Intervention): healthy volunteers

INTERVENTIONS:
Drug: prescribing anapproved drug, examination — * Blood test to assess serum zonulin levels;
  * Esophagogastroduodenoscopyand colonoscopy with biopsy from the small and large intestine followed by histological examination;
  * Stool sample collection to assess short-chain fatty acid levels and the composition of the gut microbiota.
  Then the patients were prescribed therapy with the approved drug trimebutin (trimedat) with placebo or trimebutine with rebamipide or rebamipide with placebo for 2 months.
  Other Names: Trimedate, Rebagit
  Arms: Group A; Group B; Group C

SUMMARY:
Patients with diarrhea-predominant irritable bowel syndrome (IBS) and functional dyspepsia (FD) were examined and received treatment in the study. Severity of complaints and quality of life patients were assessed according to questionnaires. The state of the intestinal barrier (analysis of the protein composition, intestinal mucin levels in biopsies, serum zonulin level in blood), the composition of the gut microbiota (16S rRNA gene sequencing), bacterial metabolic function (short-chain fatty acid levels in feces), and the presence of gut inflammation (levels of lymphocytes and eosinophils in biopsies) were assessed in the patients. Patients were divided into 3 treatment groups: trimebutin + placebo, rebamipide + placebo, trimebutin + rebamipide. The above parameters were compared in patients before and after treatment.

DETAILED DESCRIPTION:
The study included 60 patients with an established diagnosis IBS and FD. Patients were randomized in toone of three groups. Patients in group 1 received Trimedat (trimebutine, marketing authorization number LP-005534/07 of 2007-12-28) for 2 months, patients in group 2 received Trimedat and Rebagit (rebamipide, marketing authorization number LP-001831 of 2012-09-12) for 2 months, patients in group 3 received Rebagit for 2 months. The patients were blinded to the treatment assignment. At inclusion and 1 month after the severity of complaints were assessed, 2 months after starting treatment, the severity of complaints, quality of life, state of tight junction proteins, mucin-2 expression level, serum zonulin level, histological investigation of the mucous membrane of the small and large intestine, state of the intestinal microbiota and short-chain fatty acid levels were assessed. After the end of the study, an interim analysis of the effect of the therapy on the parameters was carried out. In the case of a positive effect, a full analysis of all the aforementioned factors contributing to its development was to be performed.

In addition, all these parameters were also in the control group (15 healthy volunteers without complaints, matched for sex and age with the main group).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* A man or woman aged 18-59.
* For women of childbearing age: mandatory use of contraceptive methods.
* Confirmed diagnosis of IBS-D and functional dyspepsia by clinical, instrumental and blood chemistry findings (according to the Clinical Guidelines of the Russian Gastroenterological Association and the Russian Association of Coloproctologists (2016)
* Absence of Helicobacter Pylori infection according to the urea breath test in the past 6 months before inclusion.
* Ability to understand and willingness to comply with all protocol details.

Exclusion Criteria:

* Prematurely discontinuation of the consumption of tested drugs/placebo;
* Started taking antibiotics, other probiotics, or prebiotics during the follow-up period;
* Refusal to participate during the follow-up period, including refusal to come for re-examination 2 months after inclusion;
* Cancer or inflammatory bowel disease diagnosis during the follow-up period.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Severity of complaints | change from baseline points of questionnaires at 2 months
  The severity of complaints is assessed using "7×7" (7 symptoms per 7 days) questionnaire and GSRS (Gastrointestinal Symptom Rating Scale)
Low-grade inflammation | change from baseline numbers of eosinophils and lymphocytes at 2 months
  In biopsies of the small and large intestine, numbers of eosinophils and lymphocytes in the field of view were assessed by histological examination with hematoxylin-eosin staining

SECONDARY OUTCOMES:
Tight junction protein level | change from baseline tight junction proteins levels at 2 months
  In biopsies of the small and large intestine, tight junction proteins levels are assessed by two-dimensional electrophoresis
Mucin-2 expression | change from baseline level of Mucin-2 at 2 months
  The level of Mucin-2 expression in biopsies of the small and large intestine is assessed by immunohistochemistry
Serum zonulin | change from baseline level of serum zonulin at 2 months
  The level of the permeability marker, serum zonulin, is assessed by enzyme-linked immunosorbent assay using an ELISA test kit (Immundiagnostik AG, Bensheim, Germany)
Gut microbiome | change from baseline composition of the gut microbiota in feces at 2 months
  The composition of the gut microbiota in feces is analyzed by 16S rRNA sequencing
Short-chain fatty acids | change from baseline short-chain fatty acid levels at 2 months
  Short-chain fatty acid levels in feces are assessed by gas chromatography-mass spectrometry
Adverse events | 2 months after the start of the study
  Patients are notified of the need to report any adverse and unintended signs (any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product)
Quality of life (general health, limitation of activities, physical health problems, emotional health problems, social activities, pain, energy and emotions, social activities, general health) | change from baseline points of questionnaire levels at 2 months
  Quality of life ((general health, limitation of activities, physical health problems, emotional health problems, social activities, pain, energy and emotions, social activities, general health) was assessed using the 36-Item Short Form Survey (SF-36) questionnaire
Severity of complaints | baseline
  The severity of complaints is assessed using "7×7" (7 symptoms per 7 days) questionnaire and GSRS (Gastrointestinal Symptom Rating Scale)
Low-grade inflammation | baseline
  In biopsies of the small and large intestine, numbers of eosinophils and lymphocytes in the field of view were assessed by histological examination with hematoxylin-eosin staining
Tight junction protein level | baseline
  In biopsies of the small and large intestine, tight junction proteins levels are assessed by two-dimensional electrophoresis
Mucin-2 expression | baseline
  The level of Mucin-2 expression in biopsies of the small and large intestine is assessed by immunohistochemistry
Serum zonulin | baseline
  The level of the permeability marker, serum zonulin, is assessed by enzyme-linked immunosorbent assay using an ELISA test kit (Immundiagnostik AG, Bensheim, Germany)
Gut microbiome | baseline
  The composition of the gut microbiota in feces is analyzed by 16S rRNA sequencing
Short-chain fatty acids | baseline
  Short-chain fatty acid levels in feces are assessed by gas chromatography-mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Ivashkin, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- Elena Poluektova, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
Data disclosure is not permitted by the local ethics committee. For more information about the study, please contact the principal investigator.

REFERENCES:
- [Result] Ivashkin V, Poluektov Y, Kogan E, Shifrin O, Sheptulin A, Kovaleva A, Kurbatova A, Krasnov G, Poluektova E. Disruption of the pro-inflammatory, anti-inflammatory cytokines and tight junction proteins expression, associated with changes of the composition of the gut microbiota in patients with irritable bowel syndrome. PLoS One. 2021 Jun 11;16(6):e0252930. doi: 10.1371/journal.pone.0252930. eCollection 2021. PMID 34115808
- See also: Kovaleva A.L., Poluektova E.A., Shifrin O.S. Intestinal Barrier, Permeability and Nonspecific Inflammation in Functional Gastrointestinal Disorders. Russian Journal of Gastroenterology, Hepatology, Coloproctology. 2020;30(4):52-59. (In Russ.) — https://www.gastro-j.ru/jour/article/view/437